CLINICAL TRIAL: NCT00837564
Title: Differential Responses to Cognitive Behavioural Analysis System of Psychotherapy (CBASP)Versus Escitalopram in Chronic Major Depression With and Without Early Trauma
Brief Title: Cognitive Behavioural Analysis System of Psychotherapy (CBASp) Versus Escitalopram in Chronic Depression
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Freiburg (Other)
Collaborators: University Hospital, Bonn (Other)
Responsible Party: Dr. Claus Normann, University of Freiburg, Dep. of Psychiatry, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CBASP-1
Record Dates: First submitted 2009-02-04; First posted 2009-02-05 (Estimated); Last update posted 2010-06-30 (Estimated); Status verified 2010-07

CONDITIONS: Chronic Depression
Keywords: chronic depression; CBASP; Escitalopram; depression; trauma
MeSH Terms: conditions — Depression; Wounds and Injuries | interventions — Escitalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBASP (Experimental): CBASP psychotherapy
  Interventions: Other: CBASP psychotherapy
- Escitalopram (Experimental): Escitalopram pharmacotherapy and clinical management
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Other: CBASP psychotherapy — specific psychotherapy for chronic depression
  Arms: CBASP
Drug: Escitalopram — Escitalopram 10-20 mg once daily for the treatment of depression in combination with clinical management
  Arms: Escitalopram

SUMMARY:
60 patients with chronic major depressive disorder according to DSM-IV will be included into the study. Patients will be randomized to receive an open treatment either with CBASP, a psychotherapy for chronic depression, or pharmacological treatment with Escitalopram for 28 weeks.

DETAILED DESCRIPTION:
The psychotherapeutic treatment with CBASP will be conducted in 2 weekly sessions for the first 4 weeks, one per week thereafter until week 9, followed by one session every 2 weeks for 20 more weeks. The starting dose for Escitalopram will be 10 mg/d for one week and will be increased to 20 mg/d after one week. The dosage can be reduced to 10 mg/d after day 7 to improve tolerance. Th MADRS-scale is the primary outcome measure; ratings will be performed by a blinded rater. If there is no improvement (reduction of less than 20% of the MADRS), patients will be crossed over in terms of adding the other treatment at week 8. Study patients will be asked to participate in fMRI, genetic and pharmacological substudies.

ELIGIBILITY:
Inclusion Criteria:

* Chronic MDD according to DSM-IV (modification: depressive symptomatology for at least one year), or recurrent MDE (third or greater episode with the immediately preceding episode being no more than 2.5 years before the onset of the present episode)
* Age 18-65
* Score of at least 18 on the Montgomery-Asberg-Rating Scale for Depression (MADRS)

Exclusion Criteria:

* Acute risk for suicide
* History of psychotic symptoms, bipolar disorder or dementia
* Severe substance-related abuse or dependence disorder
* Schizotypal, antisocial or borderline personality disorder
* Serious medical condition
* Severe cognitive impairment
* Absence of a response to previous adequate trial of the study medication/CBASP
* Hypersensitivity to Escitalopram
* Treatment with a MAO-inhibitor within 1 week before the initiation of study treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-02; Primary Completion 2010-04 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Depressive symptomatology after 8 weeks after randomization as measured by the MADRS | 8 weeks

SECONDARY OUTCOMES:
Depressive symptoms and remission 28 weeks after randomization; social, interpersonal and work function 28 weeks after randomization | 28 weeks after ranomization

CONTACTS AND LOCATIONS:
Overall Officials: Claus Normann, MD, Principal Investigator — University of Freiburg, Dep. of Psychiatry; Dieter Schoepf, MD, Principal Investigator — University of Bonn, Clinic for Psychiatry and Psychotherapy
Locations (2):
- Germany (2):
  - University of Bonn, Dept. of Psychiatry, Bonn
  - University of Freiburg, Dept. of Psychiatry and Psychotherapy, Freiburg im Breisgau